CLINICAL TRIAL: NCT06586554
Title: Comparative Effectiveness of Static Stretching Versus Myofascial Release on Hamstring Muscle Tightness in IT Professionals: A Randomized Comparative Study
Brief Title: Efficacy of Different Stretching Techniques on Hamstring Muscle Tightness in IT Professionals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, AMIR IQBAL, Researcher, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RRC-2020-04
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hamstring Tightness; Hamstring Flexibility
Keywords: Functional ability; Static Stretching; Myofascial Release; Hamstring tightness; Hamstring flexibility
MeSH Terms: interventions — Muscle Stretching Exercises; Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SS Group (Experimental): SS group received a static stretching on the hamstring muscle
  Interventions: Other: Static stretching
- MFR Group (Active Comparator): The MFR group received a myofascial release on the hamstring muscle
  Interventions: Other: Myofascial release

INTERVENTIONS:
Other: Static stretching — The SS group received static stretching, which was applied with gentle and firm pressure while pulling opposite the hamstring muscle contraction.
  Arms: SS Group
Other: Myofascial release — Myofascial release is applied with cross-handed stretches over hamstring muscle
  Arms: MFR Group

SUMMARY:
Brief Summary

This clinical trial aims to learn if static stretching and myofascial release work to improve hamstring muscle tightness and lower limb functional ability among IT professionals. It will also learn about the superiority of one maneuver over another. The main questions it aims to answer are:

* Does static stretching and myofascial release work to improve hamstring muscle tightness and lower limb functional ability among IT professionals?
* Which stretching maneuver is more effective in reducing hamstring muscle tightness and improving the lower limb functional ability among IT professionals? Researchers will compare static stretching to myofascial release to see if both work equally or are superior to each other in reducing hamstring muscle tightness and improving lower limb functional ability among IT professionals.

Participants will:

* Both groups received an application of hot packs for 20-25mins at the posterior aspect of the thigh.
* In addition, group 1 performed static stretching of the hamstring muscles for thirty seconds, with a thirty-second gap, repeating the same maneuver three times/day for five days/week for three weeks.
* Group 2 received a myofascial release. This maneuver involves the proper positioning of the practitioner's hands on both sides of the hamstrings, pulling them in opposite directions with firm pressure, and holding the stretch for three to five minutes each stretch, completing five to seven stretches per session with a gap of two minutes between each stretch, and continued five sessions per week for three weeks.

DETAILED DESCRIPTION:
Tightness in the hamstring muscles presents a considerable issue for many people, especially those in professions requiring long sitting periods, such as IT workers. This group often experiences a high rate of hamstring tightness because their jobs involve extended sitting and minimal physical movement. As a result, IT professionals may suffer from limited knee extension and reduced functionality, leading to discomfort and lower productivity at work and in daily activities.

The impact of hamstring tightness on knee extension and overall function has been extensively studied across various populations. Limited knee extension, commonly associated with hamstring tightness, can disrupt standard walking patterns and affect joint stability, raising the risk of musculoskeletal injuries, particularly around the knee. Additionally, the reduced functional ability caused by hamstring tightness can negatively influence daily tasks, job performance, and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* IT professionals
* males and females)
* aged between 30 and 45 years
* working in passive roles for at least 6 hours a day, and
* reported symptoms of hamstring muscle tightness such as decreased flexibility and discomfort during prolonged sitting, and found positive active knee extension test.

Exclusion Criteria:

* History of musculoskeletal injuries or neurological disorders affecting lower limb function, and
* showed non-cooperation.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Active knee extension range of motion (AKE-ROM) | 3 weeks
  Hamstring muscle tightness was assessed by active knee extension ROM using a standard full-circle goniometer. The knee angle should be between 80-90 degrees. If the range is below 80 degrees, then that subject has a tight hamstring.

SECONDARY OUTCOMES:
Lower extremity functional scale (LEFS) | 3 weeks
  Lower limb functional ability was assessed using a lower extremity functional scale. The Lower Extremity Functional Scale (LEFS) is scored on a scale of 0 to 80, with higher scores indicating better lower limb function. The interpretation of the scores can be based on the following categories: 0-20: Severe functional limitation; 21-40: Moderate functional limitation; 41-60: Mild to moderate functional limitation; 61-80: Minimal functional limitation or normal function.

CONTACTS AND LOCATIONS:
Overall Officials: AMIR IQBAL, MPT, Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Ar-Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No